CLINICAL TRIAL: NCT07367269
Title: The Effect of Mandala Coloring on Psychological Distress, Anxiety, and Comfort in Breast Cancer Patients Receiving Outpatient Chemotherapy
Brief Title: Effect of Mandala Coloring on Anxiety, Distress, and Comfort in Breast Cancer Patients Receiving Outpatient Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, EMRE ERKAL, Dr, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MANDALA-BC-CHEMO-01
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Coloring Group (Experimental): Participants will perform mandala coloring for 30 minutes during outpatient chemotherapy in addition to routine care.
  Interventions: Behavioral: Mandala Coloring
- Control group (No Intervention): Participants will receive routine outpatient chemotherapy care without any additional activity.

INTERVENTIONS:
Behavioral: Mandala Coloring — Mandala coloring activity performed for 30 minutes during outpatient chemotherapy using mandala coloring books and colored pencils.
  Arms: Mandala Coloring Group

SUMMARY:
Breast cancer patients receiving chemotherapy often experience psychological distress, anxiety, and discomfort during treatment. Non-drug supportive methods may help improve patients' well-being during chemotherapy.

This study aims to evaluate whether mandala coloring during outpatient chemotherapy can reduce psychological distress and anxiety and improve comfort in breast cancer patients. Participants will be randomly assigned to either a mandala coloring group or a routine care group. Patients in the intervention group will color mandala patterns for 30 minutes during their chemotherapy session, while the control group will receive routine care only.

Psychological distress, anxiety, and comfort levels will be measured before and after the chemotherapy session in both groups. The results of this study may provide evidence for a simple and low-cost supportive intervention to improve the psychological well-being of breast cancer patients during chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies among women and chemotherapy is a fundamental component of its treatment. However, chemotherapy is frequently associated with psychological distress, anxiety, and decreased comfort, which may negatively affect patients' quality of life and treatment adherence. Supportive non-pharmacological interventions that are easy to apply during chemotherapy are therefore needed.

Mandala coloring is a complementary approach that has been reported to reduce anxiety and psychological distress and improve well-being in patients with cancer. Nevertheless, evidence regarding its effectiveness during outpatient chemotherapy sessions remains limited. This study is designed to evaluate the effect of mandala coloring applied during outpatient chemotherapy on psychological distress, anxiety, and comfort in breast cancer patients.

This study is a randomized controlled experimental trial that will be conducted in the Chemotherapy Unit of Artvin State Hospital. A total of 60 breast cancer patients receiving outpatient chemotherapy will be recruited. Participants will be randomly assigned in a 1:1 ratio to either an intervention group (mandala coloring) or a control group (routine care). Block randomization with allocation concealment using sequentially numbered opaque sealed envelopes will be used.

Patients in the intervention group will perform mandala coloring for 30 minutes starting at the beginning of their chemotherapy session. They will be provided with mandala coloring books and colored pencils and will continue to receive routine medical care during the session. Patients in the control group will receive routine care only, without any coloring activity.

Psychological distress, anxiety, and comfort will be assessed before and after the chemotherapy session in both groups. Distress will be measured using the Distress Thermometer. Anxiety will be evaluated using the State Anxiety subscale of the State-Trait Anxiety Inventory. Comfort will be assessed using the General Comfort Scale. Pre-test and post-test measurements will be compared between groups to determine the effect of the mandala coloring intervention.

The findings of this study may contribute evidence for a simple, low-cost, and easily applicable supportive intervention to improve psychological well-being and comfort in breast cancer patients undergoing outpatient chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having a diagnosis of breast cancer and receiving chemotherapy
* Having no communication problems
* Having no physical disability that would prevent mandala coloring
* Being willing to participate in the study

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Before chemotherapy session and immediately after the chemotherapy session (single session).
  Psychological distress will be measured using the Distress Thermometer. Participants rate their level of distress on a scale from 0 (no distress) to 10 (extreme distress). Higher scores indicate greater psychological distress.

SECONDARY OUTCOMES:
Anxiety | Before chemotherapy session and immediately after the chemotherapy session (single session).
  Anxiety will be measured using the State Anxiety subscale of the State-Trait Anxiety Inventory (STAI-S). Scores range from 20 to 80, with higher scores indicating higher levels of anxiety.
Comfort | Before chemotherapy session and immediately after the chemotherapy session (single session).
  Comfort will be measured using the General Comfort Scale. Scores range from 1 to 4, with higher scores indicating higher levels of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Artvin State Hospital, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] [1] Winters S, Martin C, Murphy D, Shokar NK. Breast Cancer Epidemiology, Prevention, and Screening. Prog Mol Biol Transl Sci 2017;151: 1-32. [2] El Masri J, Phadke S. Breast Cancer Epidemiology and Contemporary Breast Cancer Care: A Review of the Literature and Clinical Applications. Clin Obstet Gynecol 2022;65: 461-481. [3] Xiong X, Zheng LW, Ding Y, Chen YF, Cai YW, Wang LP, Huang L, Liu CC, Shao ZM, Yu KD. Breast cancer: pathogenesis and treatments. Signal Transduct Target Ther 2025;10: 49. [4] Wang J, Wu SG. Breast Cancer: An Overview of Current Therapeutic Strategies, Challenge, and Perspectives. Breast Cancer (Dove Med Press) 2023;15: 721-730. [5] Bourdeanu L, Liu EA. Systemic Treatment for Breast Cancer: Chemotherapy and Biotherapy Agents. Seminars in Oncology Nursing 2015;31: 156-162. [6] Phongnopakoon P, Kongvattananon P, Somprasert C. Nursing Outcomes of Patient's Comfort during Neoplastic Chemotherapy: An Integrative Review. The Bangkok Medical Journal 2018;14: 115. [7] Oh P-J, Cho J-R. Changes in fatigue, psychological distress, and quality of life after chemotherapy in women with breast cancer: a prospective study. Cancer nursing 2020;43: E54-E60. [8] Burrai F, Sguanci M, Petrucci G, De Marinis MG, Piredda M. Effectiveness of immersive virtual reality on anxiety, fatigue and pain in patients with cancer undergoing chemotherapy: A systematic review and meta-analysis. European Journal of Oncology Nursing 2023;64: 102340. [9] Hormozi M, Hashemi SM, Shahraki S. Investigating Relationship between Pre- and Post- Chemotherapy Cognitive Performance with Levels of Depression and Anxiety in Breast Cancer Patients: A Cross-Sectional Study. Asian Pac J Cancer Prev 2019;20: 3831-3837. [10] Guo Y-Q, Ju Q-M, You M, Liu Y, Yusuf A, Soon LK. Depression, anxiety and stress among metastatic breast cancer patients on chemotherapy in China. BMC nursing 2023;22: 33. [11] Li YC, Ma SC, Wang HH. Emotional Distress in Patients With Cancer: A Cross-Sectional Study. J Nurs Res 2